CLINICAL TRIAL: NCT00247169
Title: Vaginal Progesterone in the Treatment of Cervical Dysplasia Grade I and II: A Phase II Trial
Brief Title: Vaginal Progesterone in the Treatment of Cervical Dysplasia Grade I and II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, LHefler, Assoc Professor, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFK-HEF 4
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: cervical intraepithelial neoplasia (CIN); progesterone
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Progesterone

INTERVENTIONS:
Drug: progesterone — Micronized progesterone 400mg 1x daily for 10 days/month from menstrual cycle day 16-25

SUMMARY:
The investigators want to test whether treatment with a natural progesterone intravaginally increases the cure rate of cervical intraepithelial neoplasia grade I and II.

DETAILED DESCRIPTION:
Background:

1. The development of cervical intraepithelial neoplasia (CIN) was linked to a decreased local immune response as evidenced by a decrease of Langerhans' cell (LC) count in the cervical epithelium. Preliminary studies show that vaginally administered progesterone locally increases the number of LCs.
2. There is no accepted treatment strategy of low grade CIN, i.e., CIN I and II, than await spontaneous regression.

Thus, vaginal progesterone is expected to increase the regression rate of cervical dysplasia grade I and II.

Outcome parameters:

Primary outcome parameters:

To evaluate whether or not a treatment with vaginal progesterone increases regression and remission rates of CIN I and II during a 6-month treatment period.

Secondary outcome parameters:

Change of immunohistochemically detected expression of LCs in CIN.

Methods:

Prospective phase II trial with vaginal progesterone as treatment of CIN I and II. 60 patients receive vaginal micronized progesterone 400mg 1x daily for 10 days/month from menstrual cycle day 16-25 for 6 months. After 3 and 6 months patients are examined for possible regression, persistence, or progression of disease and treated accordingly. Treatment of patients with progressing CIN is being discontinued after 3 months. Follow-up of patients is ensured based on current clinical practice, i.e., regular outpatient visits every 3 months, until the lesion completely regresses.

Diagnosis and main inclusion criteria:

CIN I and II diagnosed by punch biopsy, lesion fully visible, otherwise healthy subjects < 60 years, no history of breast cancer, patient's compliance

Medication:

Micronized progesterone 400mg 1x daily for 10 days/month from menstrual cycle day 16-25

Duration of treatment:

6 months

ELIGIBILITY:
Inclusion Criteria:

1. Histological evidence of CIN I and II
2. Transformation zone and lesion margins fully visible
3. Compliant subject
4. Safe contraception
5. Negative pregnancy test

Exclusion Criteria:

Lesion related

1. CIN III, (micro)-Invasive Cancer
2. Endocervical lesion, upper margin of lesion not visible on colposcopy
3. Non-compliance of patient
4. PAP V

Drug related

1. Age > 60
2. Hypersensitivity to progesterone or any component of the formulation
3. Thrombophlebitis
4. Undiagnosed vaginal bleeding
5. Carcinoma of the breast
6. Cerebral apoplexy
7. Severe liver dysfunction
8. Pregnancy
9. Depression
10. Diabetes
11. Epilepsy
12. Migraine
13. Renal dysfunction
14. Asthma
15. HIV infection
16. Hepatitis B or C
17. Concurrent use of anticoagulants
18. Uncontrolled hypertension (> 160/90 mmHg)
19. Breast cancer in personal history
20. Concurrent hormonal therapy including OC

Clinical laboratory related

1. Hemoglobin < 11 g/dl
2. Leukocytes < 4,0 x 109/L
3. Platelet count < 100 x 109/L
4. Serum bilirubin > 2 x above upper cut-off value
5. Serum GOT > 2 x above upper cut-off value
6. Serum GPT > 2 x above upper cut-off value
7. Serum alkaline phosphatase > 2 x above upper cut-off value
8. Serum creatinine > 2 x above cut-off value

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-08; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To evaluate whether or not a treatment with vaginal progesterone 400mg 1x daily for 10 days/month from menstrual cycle day 16-25 for 6 months increases regression rates of CIN I and II. | 6 months

SECONDARY OUTCOMES:
Change of immunohistochemically detected expression of Langerhans Cells in CIN | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lukas A Hefler, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept OB/GYN, Med University of Vienna, Vienna, Austria